CLINICAL TRIAL: NCT00494754
Title: Clinical and Genetic Study of Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 9561709027
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Autism
Keywords: autism spectrum disorder; family genetic study; gene; phenotype; endophenotype
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to prepare instruments for Autism Spectrum Disorder (ASD), to collect clinical, neuropsychological, and genetic data of ASD probands and their family, and to identify the genetic variants close to etiological genes of ASD in a Taiwanese sample

DETAILED DESCRIPTION:
Autism is a pervasive neurodevelopmental disorder with prominent reciprocal social and communication impairment and restricted repetitive behavior or interest. Based on the number of symptoms and functional impairment, autistic disorder, Asperger disorder, and atypical autism (or PDDNOS) are conceptualized as the autism spectrum disorder (ASD). Most recent survey estimated the prevalence of narrow diagnosis of autistic disorder to be around 0.1% to 0.2%, and 0.59 % to 0.63% for ASD, with a four-fold male predominance. Due to high heritability (> 0.9), high family recurrence risk (λ = 60), and severe impairment without effective prevention and treatment available for ASD, this disastrous disease has been prioritized for molecular genetic study from public health perspective. The proposed research is the first systematic approach combining clinical and molecular genetic study of ASD involving multi-sites and three research cores: assessment core (by Gau SS and Wu YY), molecular genetics core (by Chen CH), and data/statistics core (by Gau SS).

The long-term objective of this study is to establish clinical and genetic database of autism and their family for etiology study, exploration of pathogenesis, and developing new treatment. The specific aims are:

1. to establish the psychometric properties of three Chinese versions of rating scales for ASD: SCQ, SRS, and ABC;
2. to collect clinical, neuropsychological, and genetic data of ASD probands and their family and
3. to identify the genetic variants close to etiological genes of ASD in a Taiwanese sample using candidate gene case-control association study design (e.g., Neuroligin gene family, MeCP2 gene, and FOXP2 gene, parent trio and population-based studies) and whole genome linkage analysis for multiplex families.

After well-preparation of instruments, DNA collection procedure, and assessor's training in the first 6 months, we will recruit 40, 170, and 90 ASD families in the first, second, and third year of the project, respectively. The instruments include the ADI-R, ADOS, K-SADS-E, SCQ, SRS, and ABC for measuring autistic psychopathology; WISC-III, MSEL and PPVT for cognitive ability; CPT, CANTAB, and WCST for neuropsychological functioning, and MRI, MRS, and DSI for brain imaging study.

We anticipate the establishment of the database of 300 ASD families, completion of the mutation screening of several candidate genes, and determination of their association with ASD and its intermediate phenotype in our sample. The identification of susceptible genes for ASD would be a major breakthrough in child psychiatry because this revelation would facilitate the scientific diagnosis of autism and as a result, it would shed light on the pathogenesis of autism and contribute to the development of the novel, specific and effective treatment of this devastating disease.

ELIGIBILITY:
Inclusion Criteria:

1. subjects have a clinical diagnosis of autistic disorder, Asperger disorder, or atypical autism defined by the DSM-IV and ICD-10, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits;
2. their ages range from 3 to 18 when we conduct the study;
3. subjects have at least one biological parent;
4. both parents are Han Chinese; and (5) subjects and their biological parents (and siblings if any) consent to participate in this study for complete phenotype assessments and blood withdraw for genetic study

Exclusion Criteria:

1. if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, or Organic Psychosis.
2. if they completely cannot cooperate with blood withdrawal, collection of saliva, or buccal swabs.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will consist of 300 children and adolescents with ASD, aged 3-18.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (4):
- Taiwan (4):
  - National Taiwan University Hospital, Taipei
  - Taipei City Psychiatric Center, Taipei
  - Chang Gung Children's Hospital, Taoyuan District
  - Taoyuan Mental Hospital, Taoyuan District

REFERENCES:
- [Derived] Chien YL, Chen YC, Chiu YN, Tsai WC, Gau SS. A translational exploration of the effects of WNT2 variants on altered cortical structures in autism spectrum disorder. J Psychiatry Neurosci. 2021 Dec 3;46(6):E647-E658. doi: 10.1503/jpn.210022. Print 2021 Nov-Dec. PMID 34862305
- [Derived] Chien YL, Wu YY, Chen HI, Tsai WC, Chiu YN, Liu SK, Gau SS. The central nervous system patterning gene variants associated with clinical symptom severity of autism spectrum disorders. J Formos Med Assoc. 2017 Oct;116(10):755-764. doi: 10.1016/j.jfma.2016.11.015. Epub 2017 Jan 9. PMID 28081867
- [Derived] Yin CL, Chen HI, Li LH, Chien YL, Liao HM, Chou MC, Chou WJ, Tsai WC, Chiu YN, Wu YY, Lo CZ, Wu JY, Chen YT, Gau SS. Genome-wide analysis of copy number variations identifies PARK2 as a candidate gene for autism spectrum disorder. Mol Autism. 2016 Apr 1;7:23. doi: 10.1186/s13229-016-0087-7. eCollection 2016. PMID 27042285
- [Derived] Chiu YN, Chou MC, Lee JC, Wong CC, Chou WJ, Wu YY, Chien YL, Gau SS. Determinants of maternal satisfaction with diagnosis disclosure of autism. J Formos Med Assoc. 2014 Aug;113(8):540-8. doi: 10.1016/j.jfma.2012.07.040. Epub 2012 Nov 6. PMID 25037759
- [Derived] Chen CH, Huang CC, Cheng MC, Chiu YN, Tsai WC, Wu YY, Liu SK, Gau SS. Genetic analysis of GABRB3 as a candidate gene of autism spectrum disorders. Mol Autism. 2014 Jun 25;5:36. doi: 10.1186/2040-2392-5-36. eCollection 2014. PMID 24999380
- [Derived] Lau WY, Gau SS, Chiu YN, Wu YY. Autistic traits in couple dyads as a predictor of anxiety spectrum symptoms. J Autism Dev Disord. 2014 Nov;44(11):2949-63. doi: 10.1007/s10803-014-2151-5. PMID 24907095
- [Derived] Chien WH, Gau SS, Liao HM, Chiu YN, Wu YY, Huang YS, Tsai WC, Tsai HM, Chen CH. Deep exon resequencing of DLGAP2 as a candidate gene of autism spectrum disorders. Mol Autism. 2013 Aug 1;4(1):26. doi: 10.1186/2040-2392-4-26. PMID 23915500
- [Derived] Chien WH, Gau SS, Chen CH, Tsai WC, Wu YY, Chen PH, Shang CY, Chen CH. Increased gene expression of FOXP1 in patients with autism spectrum disorders. Mol Autism. 2013 Jul 1;4(1):23. doi: 10.1186/2040-2392-4-23. PMID 23815876
- [Derived] Lin PI, Chien YL, Wu YY, Chen CH, Gau SS, Huang YS, Liu SK, Tsai WC, Chiu YN. The WNT2 gene polymorphism associated with speech delay inherent to autism. Res Dev Disabil. 2012 Sep-Oct;33(5):1533-40. doi: 10.1016/j.ridd.2012.03.004. Epub 2012 Apr 21. PMID 22522212
- [Derived] Chien YL, Wu YY, Chen CH, Gau SS, Huang YS, Chien WH, Hu FC, Chao YL. Association of HLA-DRB1 alleles and neuropsychological function in autism. Psychiatr Genet. 2012 Feb;22(1):46-9. doi: 10.1097/YPG.0b013e32834915ae. PMID 21716163